CLINICAL TRIAL: NCT01246921
Title: Effect of Fluticasone Proprionate 0.05% Cream on Narrow Band UV-B Phototherapy in Active Vitiligo: a Randomised Single Blinded Controlled Trial
Brief Title: Effect of Fluticasone Proprionate 0.05% on Narrow Band UV-B in Active Vitiligo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Netherlands Institute for Pigment Disorders, Academic Medical Centre, Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNIP_UVB
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2009-06

CONDITIONS: Patients With Active Non-segmental Vitiligo.; Evaluation of the Efficacy of UVB and Fluticason Proprionate 0.05%; Cream Compared to NB-UVB Alone in Patients With Non-segmental Vitiligo
Keywords: Vitiligo, repigmentation, satisfaction
MeSH Terms: conditions — Vitiligo; Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- fluticasone proprionate 0.05 % (Active Comparator): Group reveiving 12 months NB-UVB phototherapy twice a week in combination with fluticasone proprionate 0.05 % cream in an intermittent scheme
  Interventions: Drug: Fluticasone proprionate 0.05% cream
- no intervention (No Intervention): Group receiving 12 months NB-UVB phototherapy twice weekly, without any topical treatment

INTERVENTIONS:
Drug: Fluticasone proprionate 0.05% cream — Fluticasone proprionate 0.05% cream . In each patient a representative target lesion will be selected which will be assessed by digital analysis. Patients will apply Fluticasone proprionate 0.05% cream once daily during the first 3 months. I nthe following 9 months FP will be applied in a scheme of 3 days per week
  Other Names: Cutivate cream
  Arms: fluticasone proprionate 0.05 %

SUMMARY:
Rationale: Vitiligo vulgaris is a common acquired pigment disorder, which is characterised by the development of depigmented macules. It develops probably due to immunedestruction of melanocytes. Most effective therapies are immunsuppresive:

1. local immunesuppressives like corticosteroids and calcineurin inhibitors
2. phototherapy like PUVA and NB-UVB phototherapy. NB-UVB is the first choice A synergistic effect of UVA and topical corticosteroids (fluticasone proprionate 0.05% cream) has been described by Westerhof et al. in 1999. To our knowledge to date there are no publications comparing NB-UVB combined with a topical corticosteroid and NB-UVB alone.

Objective: The objective of this study is to evaluate the clinical effects (onset and degree of repigmentation) of fluticasone proprionate 0.05% cream (thrice weekly) on NB-UVB phototherapy twice weekly for a period of 12 months.

Study design: Prospective single blinded randomised controlled study. Study population: Consecutive patients ≥ 18 years, diagnosed with active vitiligo vulgaris who will receive NB-UVB phototherapeutic treatment at the Netherlands Institute for Pigment Disorders at the Academic Medical Centre (AMC), University of Amsterdam.

Methods: The patient will be randomised for either NB-UVB phototherapy and fluticasone proprionate 0.05% cream or NB-UVB phototherapy alone for 12 consecutive months.

Main study parameters/endpoints: The onset and degree of repigmentation is assessed by digital image analysis of a target lesion and blinded global physician assessment. Furthermore, the patients and doctors satisfaction will be assessed and changes of immunohistochemical parameters will be analysed in skin biopsies.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects participating in the study will be asked to visit the institute 4 times. The time investment will be 20 minutes per visit. Additionally, patients will be asked for consent to take punch biopsies (3 mm) at the beginning and at the end of the treatment period. Hence, skin biopsies are not compulsory for participation in this study. Patients may chose to participate in the clinical non invasive part of the study. Known side effects of the NB-UVB phototherapy are redness, pruritus, xerosis cutis, burning sensation and conjunctivitis. These side-effects however, are largely dose-dependent and avoidable. Corticosteroid associated systemic side-effects (suppression of the adrenocortex) will be minimized by treating only a limited body surface [a maximum of 30% body surface] and by using an intermittent application scheme of three days a week in the long term treatment. The regions which are known to have a higher absorption are excluded (periorbital, axillary, inguinal and genital area). Both topical corticosteroids and NB-UVB are part of the Dutch and British guidelines for the treatment of vitiligo. There is no presumptive evidence or indication that the combination of these therapies may result in a higher risk of side effects.

All together the burden due to the study is low and the risk for systemic or local side effects is low.

ELIGIBILITY:
Inclusion Criteria:

* non-segmental vitiligo
* Eligible for NB-UVB therapy
* Subjects attending the outpatient department of the SNIP
* patients > 18 years
* Skin type II-V
* patients with active vitiligo: progression of older lesions or development of new lesion during the last 6 months
* Subject is willing and able to give written informed consent

Exclusion Criteria:

* Personal or a family history of skin cancer ( non-melanoma skincancer: first degree family members, melanoma: any family members)
* Personal history of photosensitivity and/or phototoxicity disorders
* pregnancy
* Taking medication known to cause photosensitivity, phototoxicity, immune suppression and chronic or very frequent use of any medication that can influence the UVB response (e.g. tetracycline, retinoids, sulfonamids, psoralens)
* Other skin diseases that would impair the evaluation of repigmentation
* not able to have 2 times weekly NB-UVB phototherapy
* With local immunosuppressive treatment or 6 weeks prior to enrolment. For these patients a washout period of 6 weeks will be required.
* Contact-allergy for any of the parts in fluticasone proprionate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Repigmentation of the vitiligo lesions | 15 months
  Degree of repigmentation is assessed by digital analysis of a target lesion by a blinded global physician assessment

SECONDARY OUTCOMES:
Patients satisfaction | 15 months
  satisfaction/preference

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands Institute for Pigments Disorders, Amsterdam, Netherlands